CLINICAL TRIAL: NCT00370942
Title: GW823093 Japan Phase IIa Mono
Brief Title: GW823093C For The Treatment Of Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety issue
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPB106652
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GW823093C; diabetes; type 2 diabetes mellitus; DPP-IV inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- GW823093C A (Placebo Comparator): A=45 mg
  Interventions: Drug: GW823093C A
- GW823093C B (Placebo Comparator): B=30 mg
  Interventions: Drug: GW823093C B
- GW823093C C (Placebo Comparator): C=15 mg
  Interventions: Drug: GW823093C C

INTERVENTIONS:
Drug: GW823093C A — A=45 mg
  Arms: GW823093C A
Drug: GW823093C B — B=30 mg
  Arms: GW823093C B
Drug: GW823093C C — C=25 mg
  Arms: GW823093C C

SUMMARY:
This study was designed to find dose response and as extension in treatment of GW823093C.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus.
* Managed by diet therapy or receiving treatment with oral anti-diabetic monotherapy (excluding TZD (Thiazolidinediones))

Exclusion criteria:

* Patients who have metabolic disease judged by investigator as a clinically significance
* Serious cardiovascular disease or serious hepatic disease

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-04-01; Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-25 (Actual)

PRIMARY OUTCOMES:
Efficacy variables Dose response (change from baseline in HbA1c) at stipulated date in each treatment group | 12 weeks

SECONDARY OUTCOMES:
Long term safety variables | 64 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (3):
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site